CLINICAL TRIAL: NCT05869409
Title: The Relationships Between Physical Activity, Psychopathological Symptoms, and Health-Related Quality of Life in People Diagnosed With Psychotic or Affective Disorders
Brief Title: Physical Activity, Psychopathology, and Quality of Life in People With Psychotic or Affective Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Social Sciences and Humanities, Warsaw (Other)
Responsible Party: Sponsor
Other Study IDs: SWPS_01/P/01/2020
Record Dates: First submitted 2023-05-09; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Psychotic Disorders; Affective Disorder
Keywords: Physical Activity; Quality of Life
MeSH Terms: conditions — Psychotic Disorders; Mood Disorders; Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People diagnosed with a psychotic disorder or an affective disorder
  Interventions: Behavioral: Physical activity and sedentary behavior education

INTERVENTIONS:
Behavioral: Physical activity and sedentary behavior education — Enrolled patients will participate in an individual face-to-face education session, addressing: definitions and examples of sedentary and physical activity behaviors; physical health-related and mental health-related consequences of these behaviors; ways to break sedentary behaviors; age-adjusted physical activity recommendations (based on the guidelines of the World Health Organization).

SUMMARY:
This longitudinal observational study tests the associations between physical activity, health-related quality of life, and psychopathology symptoms among people diagnosed with schizophrenia or diagnosed with affective disorders. It was assumed that higher levels of physical activity at baseline will be related to better quality of life (across physical, social, and psychological domains), and lower psychopathology symptoms (positive and negative symptoms of psychosis, general psychopathology, and depression severity) at 6-week follow-up measurement. Adult participants with a diagnosis of a psychotic disorder or a diagnosis of an affective disorder will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

- a diagnosis of a psychotic disorder or affective disorder

Exclusion Criteria:

* major cognitive deficits, indicated by total scores > 8 points, obtained with the Montreal Cognitive Assessment (MoCA) Scale at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People who are participating in rehabilitation programs for individuals diagnosed with psychosis and/or affective disorders will be recruited in out-patient rehabilitation clinics. Patients treated at with pharmacotherapy and/or psychotherapy for individuals diagnosed with psychosis and/or affective disorders will be recruited in out-patient clinics.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Health-Related Quality of Life | change from the baseline health-related quality of life at 6 weeks
  scores (range 0-100) obtained in the World Health Organization Quality of Life Questionnaire (WHOQOL-BREF); higher scores indicate better quality of life

SECONDARY OUTCOMES:
Positive Symptoms (Psychosis) | change from the baseline positive symptoms at 6 weeks
  scores obtained with Positive and Negative Syndrome Scales (PANSS): Positive Symptoms subscale, scores range: 7-49; higher scores indicate more symptoms
Negative Symptoms (Psychosis) | change from the baseline negative symptoms at 6 weeks
  scores obtained with Positive and Negative Syndrome Scales (PANSS): Negative Symptoms subcale, scores range: 7-49, higher scores indicate more symptoms
General Psychopathology Symptoms )Psychosis) | change from the baseline general psychopathology symptoms at 6 weeks
  scores obtained with Positive and Negative Syndrome Scales (PANSS): General Psychopathology subscale, scores range: 16-112, higher symptoms indicate more symptoms
Depression symptoms | change from baseline depression symptoms at 6 weeks
  scores obtained in Patient Health Questionnaire -9 (PHQ-9); scores range: 0-36; higher scores indicate more severe symptoms of depression
Physical activity | change from baseline physical activity at 6 weeks
  minutes of physical activity per week measured with International Physical Activity Questionnaire - Short Form (IPAQ-Short Form); more minutes indicate more time spent on light, moderate, or high-intensity physical activity

CONTACTS AND LOCATIONS:
Locations (1):
- SWPS University, Faculty of Psychology in Wroclaw, Wroclaw, Lower Silezia, Poland

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be made open and deposited at Open Science Framework repository. Anonymized data will include aggregated (sum) scores for all outcome measures.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After data exploitation by the researchers involved in data collection.

REFERENCES:
- [Background] Development of the World Health Organization WHOQOL-BREF quality of life assessment. The WHOQOL Group. Psychol Med. 1998 May;28(3):551-8. doi: 10.1017/s0033291798006667. PMID 9626712
- [Background] Levis B, Benedetti A, Thombs BD; DEPRESsion Screening Data (DEPRESSD) Collaboration. Accuracy of Patient Health Questionnaire-9 (PHQ-9) for screening to detect major depression: individual participant data meta-analysis. BMJ. 2019 Apr 9;365:l1476. doi: 10.1136/bmj.l1476. PMID 30967483
- [Background] Kay SR, Fiszbein A, Opler LA. The positive and negative syndrome scale (PANSS) for schizophrenia. Schizophr Bull. 1987;13(2):261-76. doi: 10.1093/schbul/13.2.261. PMID 3616518
- [Background] Lee PH, Macfarlane DJ, Lam TH, Stewart SM. Validity of the International Physical Activity Questionnaire Short Form (IPAQ-SF): a systematic review. Int J Behav Nutr Phys Act. 2011 Oct 21;8:115. doi: 10.1186/1479-5868-8-115. PMID 22018588